CLINICAL TRIAL: NCT00630461
Title: Safety Study of 20,000 EU of Clinical Center Reference Endotoxin in Allergic Adults With and Without Mild Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Data collected under different protocol; funding exhuasted
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, David B. Peden, MD, Professor of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-2026 GCRC 2627
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-10

CONDITIONS: Mild Allergic Rhinitis; Mild Allergic Rhinitis With Mild Asthma
Keywords: mild asthma, mild allergies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Clinical Center Reference Endotoxin — single inhalation challenge

SUMMARY:
Endotoxin is a component of outdoor air pollution, an air contaminant found in a number of different workplaces, and is even found in homes. The endotoxin used for this study is obtained from the National Institutes of Health, and is called "Clinical Center Reference Endotoxin", or CCRE. The purpose of this Phase 1 research study is to identify a dose of inhaled endotoxin that is safe (does not cause prolonged cough, shortness of breath or other problems), but causes changes in your sputum cell samples that the scientists can measure. Phase 1 research studies like this one are not intended to be a treatment, but are a scientific investigation. Eventually, with these types of studies we will be able to examine why some people are more sensitive to endotoxin. Scientists at other universities have found that while most people do not have a considerable lung response to endotoxin at doses as high as 60,000 EU (endotoxin units), a few respond to as little as a total dose of 4500 EU. Our study is designed to identify if using a dose of 20,000 EU causes changes in the lung cells but does not cause symptoms in our study subjects. In our previous studies in our lab, using an endotoxin from another source, we have used higher doses (15,000 EUs) in subjects with asthma with no major problems, and we have used 10,000 EUs of CCRE in subjects with allergies and asthma without problems. We have used 20,000 EUs of CCRE in healthy individuals with no major problems.

ELIGIBILITY:
Inclusion Criteria:

* Mild allergic rhinitis
* Mild allergic asthma
* Normal lung function
* No other chronic illness

Exclusion Criteria:

* Use of inhaled or oral steroids
* Emergency treatment of asthma in last year
* Inhaled tobacco use

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2008-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Increased sputum neutrophils with no adverse events | 6 hours post challenge

CONTACTS AND LOCATIONS:
Overall Officials: David b Peden, MD, MS, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States